CLINICAL TRIAL: NCT03128918
Title: Non-invasive Diagnosis of Non-alcoholic Steatohepatitis in Liver Transplant Recipients: a Prospective, Longitudinal Study Employing Serum Cytokeratin 18 and Transient Elastography (Fibroscan)
Brief Title: Non-invasive Diagnosis of Non-alcoholic Steatohepatitis in Liver Transplant Recipients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Canadian National Transplant Research Program (Other)
Responsible Party: Principal Investigator, Giada Sebastiani, md, McGill University Health Centre/Research Institute of the McGill University Health Centre
Other Study IDs: 15-002-MUHC
Record Dates: First submitted 2015-08-07; First posted 2017-04-25 (Actual); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Non-alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is is to use non-invasive diagnostic tests, Fibroscan and a simple blood test, to diagnose NASH in patients who undergo liver transplantation. Liver transplantation is a life-saving procedure for people with cirrhosis. Fatty liver is a common reason for liver transplantation due to obesity and diabetes. Fatty liver can happen again to the new transplanted liver and it is often due to metabolic risk factors (including diabetes, rapid weight gain, and immunosuppressive therapy, which are used to avoid rejection of the new liver). Some patients with fatty liver after liver transplant have non-alcoholic steatohepatitis (NASH) injury to liver the tissue (inflammation) and damage which is caused by a build-up of fat in the liver. This is a serious problem and can lead to cirrhosis and loss of the transplanted liver. There has been no detailed study into the recurrence of NASH. One reason for this is one of the only ways to detect fatty liver and NASH is to have a liver biopsy, which can be painful and have complications. Recently, a new technology (Fibroscan) and a simple blood test (cytokeratin 18) have been developed which can tell doctors how much a liver is damaged and how much fat it contains without pain or complications. This is a year long study involving one screening visit and 3 study visits, 3 months apart.

DETAILED DESCRIPTION:
This is a prospective, longitudinal, pilot study of non-invasive diagnostic tests to explore recurrent or de novo NAFLD/NASH in liver transplant recipients. The study will be conducted at the Royal Victoria Hospital, McGill University Health Centre (MUHC) Solid Organ Transplant Unit, which carries out 60 liver transplants per year. A dedicated liver transplant database is in place since 1990 and prospectively collects demographic and clinical characteristics of all patients. In November 2013, two fully equipped Fibroscan machines have been acquired by the Division of Gastroenterology and Hepatology of the MUHC. The MUHC is the first center in Quebec to have access to the latest modules of Fibroscan (CAP and XL probe) that are essential to diagnose hepatic steatosis. In preparation for the current project, the Investigators performed an analysis of frequencies of hepatitis C, alcoholic liver disease, NASH, hepatitis B as indications for liver transplantation MUHC Center Solid Organ Transplant in 2000 and 2013. NASH was the only indication that significantly increased (8% in 2000 vs 20% in 2013; p<0.0001) and currently represents the third indication.

Enrolled participants will be followed every 3 months for one year, in conjunction with their regular care visit.

Blood samples obtained during the screening and the study visits will be processed by the research technician of the MUHC Solid Organ Transplant Unit. The plasma will be stored at -80C until used for quantitative measurement of CK-18 levels by the Human cytokeratin ELISA kit.

The fibroscan examination will be performed on a 4-hour fasting participants. The standard M probe will be used in all participants. The XL probe will be used in obese patients (BMI>30 Kg/m2) and in case of failure of Fibroscan by the M probe. CAP examination will be performed at the same time to diagnose hepatic steatosis. A valid Fibroscan result will be defined by 10 validated measures and IQR < 30% of the median. Validated cut-off values will be applied to diagnose hepatic steatosis and fibrosis by Fibroscan/CAP. Grading of steatosis will be as following: mild steatosis (<30% of the hepatocytes); moderate steatosis (30-60%); severe steatosis (>60%).

ELIGIBILITY:
Inclusion Criteria:

* Liver transplant recipient of any etiology;
* >18 years old;
* Able to provide informed consent.

Exclusion Criteria:

* Liver transplant due to alcoholic liver disease as primary etiology;
* Liver transplant due to chronic hepatitis C, genotype 3.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: post liver transplant
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2015-07; Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of NASH in liver transplant recipients | 18 months
  CK-18 to indicate NASH
Evaluation of liver steatosis in liver transplant recipients | 18 months
  Fibroscan with CAP to indicate steatosis
Incidence of fibrosis | 18 months
  Liver stiffness measurement by Fibroscan

SECONDARY OUTCOMES:
Accuracy of noninvasive tests to diagnose NAFLD/NASH and hepatic fibrosis as compared to standard of care histology | 18 months
  Evaluate the accuracy of CK-18 and Fibroscan/CAP

CONTACTS AND LOCATIONS:
Overall Officials: Giada Sebastiani, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- Mcgill University Health Center, Montreal, Quebec, Canada